CLINICAL TRIAL: NCT06955663
Title: Exercise Support and Rehabilitation for Patients After Spontaneous Coronary Artery Dissection- a Feasibility Study
Brief Title: Exercise Support and Rehabilitation for Patients After Spontaneous Coronary Artery Dissection
Acronym: EXERCISE-SCAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other); Edinburgh Napier University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1018; SCOT23-100002 (Other Grant/Funding Number: Heart Research UK)
Record Dates: First submitted 2025-04-15; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Spontaneous Coronary Artery Dissection
Keywords: Sponaneous coronary artery dissection; Exercise; Randomised controlled trial; Rehabilitaiton; Fesability
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: External collaborators
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): 12 week exercise intervention, + cardiopulmonary exercise test (CPET) + wearable activity monitor for the intervention period
  Interventions: Behavioral: Exercise training
- Usual care (No Intervention): Usual car + blinded activity monitor

INTERVENTIONS:
Behavioral: Exercise training — 12 week exercise intervention + cardiopulmonary exercise test (CPET) + wearable activity monitor
  Arms: Exercise Intervention

SUMMARY:
The study aims to examine the feasibility of a remote exercise program in women recovering from spontaneous coronary artery dissection (SCAD) events (heart attacks). Heart attacks caused by SCAD are different to the traditional heart attacks. In SCAD a tear happens within the blood vessels causing partial or full blockage. The population affected by SCAD is hugely different to the population affected by other 'traditional' heart attacks; as SCAD mainly happens in otherwise healthy women. From historical cases, SCAD has been associated with strenuous exercise, however, medical research did not find a link. The recovery after SCAD is also very different from other 'traditional' heart attacks. Cardiac rehab programmes are designed for an older population therefore they may not be suitable for a younger predominantly female population. This study will examine if a remote-exercise programme is achievable in people after a SCAD event.

DETAILED DESCRIPTION:
Spontaneous coronary artery dissection (SCAD) is a rare condition that leads to myocardial infraction (MI). Young women make up 87-95% of SCAD events, which is also the leading cause of MIs occurring after pregnancy. Following any MI event, cardiovascular rehabilitation (CR) is recommended, which includes supervised exercise sessions, and interventions to reduce risk factors, improve psychosocial wellbeing, and increase medication adherence. Evidence from randomised controlled trials (RCTs) show that CR reduces cardiac events and decreases mortality but this evidence is largely generated in a population with atherosclerotic disease. Trials of CR include mostly male participants, typically aged in their mid-sixties therefore CR guidelines may not be appropriate for the SCAD population who significantly differ in pathophysiology, age and gender compared with the population for which CR has been developed and tested.

Previous observational data suggested an association with strenuous exercise and SCAD, however, no casual link has been established. Clinical advice on exercise following SCAD is conflicting due to the lack of RCTs and therefore evidence. Consequently, many SCAD patients experience psychological distress, fear, and anxiety about exercise, avoiding all exercise which may lead to predictable long-term health consequences. Well-tested recovery programmes in SCAD are required to offer informed and tested exercise-based support to reduce the fear and hesitancy that may lead to exercise avoidance. This is particularly needed for women, who constitute the majority of SCAD diagnoses but are less likely to be referred to, attend, or adhere to CR. Small studies have explored the feasibility of SCAD survivors' participation in CR , however, programmes in these studies used conservative guidance preventing participants to reach pre-morbid exercise levels. This is problematic as (a) if participants are asked to exercise at levels well below their functional capacity, a rehabilitation effect is unlikely (b) such advice potentially reinforces that only lower levels of exercise are safe. This highlights the challenges SCAD survivors have in knowing what is safe and effective in terms of exercise. Therefore, this project aims to improve what we know about exercise and physical activity after SCAD.

The investigators will aim to test if women who have survived a SCAD will take part in a two-arm feasibility randomised controlled study of a 12-week remote exercise programme, what levels of exercise duration and intensity they achieve, and what they think about it. The two-arm design (usual care + blinded wearable activity monitor [control] and exercise intervention, + cardiopulmonary exercise test(CPET), + wearable activity monitor [intervention]) has been chosen to allow for the use of CPET at baseline to ensure safe exercise prescription.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged ≥18 years.
* Diagnosed with angiographically confirmed SCAD and referred to the Leicester SCAD clinic.
* Ejection fraction >45%.
* Blood pressure <180/100. Resting heart rate <100bpm

Exclusion Criteria:

* No SCAD diagnosis.
* Unable to travel to Leicester Hospital for their SCAD clinic appointment.
* Unable to give informed consent.
* No smart phone or internet access
* Unable to understand verbal explanations in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From initial patient identification until the patient consents to be part of the study. This may take up to 14 days (from initial approach until full informed consent is obtained).
  Rate of successful recruitment
Adherence | At week 8 (56 days) of the intervention.
  Rate of successful adherence
Acceptability | At 24 (168 days) of the intervention (this is follow up time point three (T3)).
  Acceptability of the intervention assessed via qualitative interviews which will be then transcribed verbatim. Acceptability will be assessed via thematic analysis of semi-structured interviews. Once patients completed T3 (+/- 7 days), they will be invited to take part in semi-structured interviews.
Signal of efficacy: Changes in exercise duration | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Changes in exercise duration expressed in time (hours: minutes) measured by the activity monitor(s) over the study period.
Signal of efficacy: Changes in exercise intensity | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Changes in exercise intensity expressed in period(s) of time spent (hours: minutes) performing light, moderate, and/or heavy intensity exercise.

SECONDARY OUTCOMES:
Self-efficacy: Self-efficacy questionnaire | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Self-reported self-efficacy levels via the self-efficacy questionnaire. This questionnaire uses a 10-item Likert scale, where minimum score is 1 (not at all true) and the maximum score is 4 (exactly true). The overall score range therefore is 10-40 where higher scores indicate better self-efficacy.
Chest pain: Seattle Angina Questionnaire-7 | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Self-reported chest pain via the Seattle Angina Questionnaire-7 (SAQ-7) uses a four week recall period therefore the scores can be translated into frequency of angina symptoms 0-30=daily angina, 31-60=weekly angina, 61-99=monthly angina and 100=no angina). The summary score range from 0 to 100 with higher scores indicating less angina and overall better quality of life.
Wellbeing: Warwick Edinburgh Mental Wellbeing Scale | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Self-reported wellbeing via the Warwick Edinburgh Mental Wellbeing Scale (WEMWBS). This is a 14-item Likert scale questionnaire with 5 response categories (1=None of the time to 5=All of the time). The total score can range from 14-70, where higher scores indicate better wellbeing.
Anxiety: Generalised Anxiety Disorder | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Self-reported general anxiety levels will be assessed via the Generalised Anxiety Disorder questionnaire (GAD-7). The GAD-7 scores each item in a Likert-scale fashion, where 'Not at all' is scored as '0', 'Several days in scored as '1' , 'More than half the days' is scored as '2' and 'Nearly every day' is scored as '3'. Higher values indicate more severe anxiety (where maximum score is 21). The data then can be categorised into the following:
  Score 0-4: Minimal Anxiety Score 5-9: Mild Anxiety Score 10-14: Moderate Anxiety Score greater than 15: Severe Anxiety.
Anxiety: Cardiac Anxiety Questionnaire | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Self-reported cardiac related questionnaire, which assesses cardiac anxiety via 18 items in a Likert-scale fashion. Items are scored from 0-4 where 'Never' is scored as '0', 'Rarely' is scored as '1' , 'Sometimes' is scored as '2' , 'Often' is scored as '3' and 'Always' is scored as '4'. Higher scores indicate more severe anxiety where the minimum score is 0 and the maximum is 72.
Demographic and health data: Age | At baseline/Day 1 (T1).
  Age expressed in years
Demographic and health data: Sex | At baseline/Day 1 (T1).
  Sex assigned at birth expressed as: Female, Male or Prefer not to answer.
Demographic and health data: Ethnicity | At baseline/Day 1 (T1).
  Categorical self-reported data defined as the following:
  * White
  * Gypsy or Irish Traveller
  * White and Black Caribbean
  * White and Black African
  * White and Asian
  * Indian
  * Pakistani
  * Bangladeshi
  * Chinese
  * African
  * Caribbean
  * Arab
  * Any other ethnic group (please describe)
  * Prefer not to answer.
Demographic and health data: Number of Spontaneous Coronary Dissection (SCAD) events | At baseline/Day 1 (T1).
  Self-reported numbers of Spontaneous Coronary Dissection (SCAD) events.
Demographic and health data: Smoking status | At baseline/Day 1 (T1).
  Self-reported smoking status defined as 'Current smoker', 'Previous smoker' and/or 'Never smoked'
Physical activity: International Physical Activity Questionnaire - short version | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Self-reported measure of momentary physical activity levels. Participants are asked to recall habitual physical activity levels (of all intensities such as vigorous, moderate activities and walking) from the past 7 days. Participants are requested to quantify time spent performing these activities in days, hours and minutes. Participants are also asked to report on sedentary time. A finals scores is then calculated and expressed in the metabolic equivalent of task (MET) minutes per week (MET/min/week).
Physical function: 6 Minute Walk Test | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Self-reported distance achieved in the 6-minute walk test administered using the Timed Walk App. Participants are requested the distance (in metres) they walked over 6 minutes.
Physical function: Sit to stand test | At week 1 (T1) of the intervention and at the end of the intervention at week 12 (T2) and at follow up of week 24 (T3).
  Participants are requested to report the number of repetitions (count data) of sit to stands over half a minute (30 seconds).

CONTACTS AND LOCATIONS:
Overall Officials: David Adlam, BA BM BCh DPhil FRCP FESC, Principal Investigator — University of Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a single site feasibility study as such we aim to gather a relatively small amount of data at one hospital site within the UK. The Principal Investigator of the study is the same medical doctor as the Principal Investigator at the hospital site therefore it is unlikely that IPD will need to be shared. Pseudonymised datasets may be shared with collaborating partners in the future.

REFERENCES:
- [Background] Hanson CL, Kelly P, Neubeck L, Bell J, Gibb H, Jin K. The Contribution of Leisure Center Usage to Physical Activity in the United Kingdom: Evidence From a Large Population-Based Cohort. J Phys Act Health. 2021 Mar 3;18(4):382-390. doi: 10.1123/jpah.2020-0422. Print 2021 Apr 1. PMID 33657530
- [Background] Neubeck L, McHale S, Ross M, MacGillivray S, Galbraith M, Hanson C. Spontaneous coronary artery dissection: a systematic review of physical and psychosocial recovery following discharge from hospital. Eur J Cardiovasc Nurs. 2022 Oct 14;21(7):665-676. doi: 10.1093/eurjcn/zvac009. PMID 35290455
- [Background] Silber TC, Tweet MS, Bowman MJ, Hayes SN, Squires RW. Cardiac rehabilitation after spontaneous coronary artery dissection. J Cardiopulm Rehabil Prev. 2015 Sep-Oct;35(5):328-33. doi: 10.1097/HCR.0000000000000111. PMID 25730096
- [Background] Imran H, Gaw A, Stabile L, Shah N, Choudhary G, Wu WC. Safety and Outcomes of Cardiac Rehabilitation for Patients with Spontaneous Coronary Artery Dissection. J Rehabil Med Clin Commun. 2018 May 23;1:1000001. doi: 10.2340/20030711-1000001. eCollection 2018. PMID 33884107
- [Background] Chou AY, Prakash R, Rajala J, Birnie T, Isserow S, Taylor CM, Ignaszewski A, Chan S, Starovoytov A, Saw J. The First Dedicated Cardiac Rehabilitation Program for Patients With Spontaneous Coronary Artery Dissection: Description and Initial Results. Can J Cardiol. 2016 Apr;32(4):554-60. doi: 10.1016/j.cjca.2016.01.009. Epub 2016 Jan 18. PMID 26923234
- [Background] Sawan MA, Calhoun AE, Fatade YA, Wenger NK. Cardiac rehabilitation in women, challenges and opportunities. Prog Cardiovasc Dis. 2022 Jan-Feb;70:111-118. doi: 10.1016/j.pcad.2022.01.007. Epub 2022 Feb 10. PMID 35150655
- [Background] Supervia M, Medina-Inojosa JR, Yeung C, Lopez-Jimenez F, Squires RW, Perez-Terzic CM, Brewer LC, Leth SE, Thomas RJ. Cardiac Rehabilitation for Women: A Systematic Review of Barriers and Solutions. Mayo Clin Proc. 2017 Mar 13:S0025-6196(17)30026-5. doi: 10.1016/j.mayocp.2017.01.002. Online ahead of print. PMID 28365100
- [Background] Binnie K, Neubeck L, McHale S, Hanson CL. What do spontaneous coronary artery dissection survivors want to support their recovery? a qualitative study. Eur J Cardiovasc Nurs. 2023 Dec 14;22(8):814-823. doi: 10.1093/eurjcn/zvad013. PMID 36656922
- [Background] Bouchard K, Tarannum CN, Coutinho T, So D, Tulloch H. Secondary Preventative Care for Patients After Spontaneous Coronary Artery Dissection: A Qualitative Analysis of Health Care Providers' Perspectives. Can J Cardiol. 2020 Jul;36(7):1156-1160. doi: 10.1016/j.cjca.2019.11.004. Epub 2019 Nov 11. PMID 32247705
- [Background] Bouchard K, Coutinho T, Reed J, Lalande K, Tarannum CN, So D, Saw J, Mulvagh S, Tulloch H. Recovering from spontaneous coronary artery dissection: Patient-reported challenges and rehabilitative intervention needs. Health Psychol. 2021 Jul;40(7):472-479. doi: 10.1037/hea0001086. PMID 34435799
- [Background] Saw J, Aymong E, Sedlak T, Buller CE, Starovoytov A, Ricci D, Robinson S, Vuurmans T, Gao M, Humphries K, Mancini GB. Spontaneous coronary artery dissection: association with predisposing arteriopathies and precipitating stressors and cardiovascular outcomes. Circ Cardiovasc Interv. 2014 Oct;7(5):645-55. doi: 10.1161/CIRCINTERVENTIONS.114.001760. Epub 2014 Oct 7. PMID 25294399
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Angelantonio ED, Franco OH, Halvorsen S, Richard Hobbs FD, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice: Developed by the Task Force for cardiovascular disease prevention in clinical practice with representatives of the European Society of Cardiology and 12 medical societies With the special contribution of the European Association of Preventive Cardiology (EAPC). Rev Esp Cardiol (Engl Ed). 2022 May;75(5):429. doi: 10.1016/j.rec.2022.04.003. No abstract available. English, Spanish. PMID 35525570